CLINICAL TRIAL: NCT02396082
Title: MIND: An RCT of Care Coordination for Community-living Person With Dementia
Brief Title: MIND: Care Coordination for Community-living Person With Dementia
Acronym: MIND at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Thomas Jefferson University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00041744; 90059611 (Other: Other); 1R01AG046274-01A1 (NIH)
Record Dates: First submitted 2015-03-10; First posted 2015-03-24 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Dementia; Caregiver Burden
Keywords: care coordination; quality of life; community-based; care quality; Long term care placement; memory care; Neuropsychiatric behaviors
MeSH Terms: conditions — Dementia; Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MIND-S Intervention (Experimental): Participants (persons with dementia (PWD) and their family caregiver (CG)) in this group will receive up to 18 months of the MIND-S dementia care coordination intervention by an interdisciplinary team comprised of trained memory care coordinators (non-clinical), a psychiatric nurse, and geriatric psychiatrist. The intervention involves 4 key components: identification of needs and individualized care planning (PWD and CG needs); dementia education and skill building; coordination, referral and linkage of services; and care monitoring.
  Interventions: Behavioral: MIND-S Intervention
- Augmented Usual Care (Other): Participants (persons with dementia (PWD) and their family caregiver (CG)) and their primary care physicians in this group will receive an initial in-home needs assessment and then a written report indicating any unmet care needs identified and potential recommendations of care for meeting those needs. They will be able to pursue any interventions or treatments they or their treating physicians deem appropriate. They will also receive a standardized Aging and Caregiver Resource Guide developed in the previous MIND trial. The study team will perform another in-home needs assessment at 18 months and the written report along with recommendations for care will be provided to the family and the PWD's primary care physician.
  Interventions: Other: Augmented Usual Care

INTERVENTIONS:
Behavioral: MIND-S Intervention — MIND at Home is a home-based, care coordination that focuses on persons with dementia living at home and their family caregivers. Its goal is to help persons age in place safely while increasing quality of life. Delivered over 18 months, MIND systematically assesses and addresses unmet care needs of persons with dementia and their caregivers which are known to be linked to poor health and quality of life outcomes, and that put people at risk for long term care placement. The needs addressed in the MIND program cover a wide range of care domains, ranging from home and medication safety, to cognitive and behavior symptoms management, meaningful activities and legal considerations. The care team made up of a memory care coordinator, nurse, and physician. Patients and families receive care coordination assistance, resource referrals, dementia care education and behavior management skills training, emotional support and problem-solving, and home safety education
  Other Names: MIND at Home - Streamlined
  Arms: MIND-S Intervention
Other: Augmented Usual Care — Augmented usual care consists of an initial full in-home needs assessment for dementia-related needs and a written report that identifies unmet needs and provides recommendations for care sent to the participant and the primary care physician. Augmented usual care participants also receive an Aging and Caregiver Resource Guide that includes program and contact information for several local and national aging service organizations (e.g., Alzheimer's Association, Administration on Aging, Centers for Medicare and Medicaid). This condition likely exceeds the usual level of intervention in primary care settings
  Arms: Augmented Usual Care

SUMMARY:
This is a 24-month, prospective, single- blind, randomized controlled trial evaluating the MIND at Home-streamlined dementia care coordination intervention (called MIND-S) in a cohort of 300 community-living persons with dementia and their family caregivers in the Greater Baltimore area. Participants receiving MIND-S will get 18 months of care coordination by an interdisciplinary team comprised of trained memory care coordinators (non-clinical), a psychiatric nurse, and geriatric psychiatrist. The intervention involves 4 key components: identification of needs and individualized care planning (persons with dementia (PWD) and care giver (CG) needs); dementia education and skill building; coordination, referral and linkage of services; and care monitoring.Participants in the comparison group will receive an initial in-home needs assessment and will be given the written results along with any recommendations for care that are indicated.

DETAILED DESCRIPTION:
Over 5 million older Americans currently suffer from Alzheimer's disease and related dementias with 80% receiving care in the community by 15 million informal caregivers (CGs) providing unpaid care. Dementia is associated with high health care costs, long term care (LTC) placement, medical complications, reduced quality of life, and CG burden. Patient and family centric care models tailored to dementia that address the multidimensional aspects of dementia management, and link health and community care are understudied but may represent a promising mechanism to address the multiple and on-going needs of this growing population, reduce adverse outcomes such as premature LTC placement, and produce cost benefits.

This is a definitive Phase III efficacy trial to test Maximizing Independence at Home-Streamlined (MIND-S), a home- based, care coordination intervention for community-living persons with dementia (PWD) and their family CGs that builds on pilot work. In a pilot trial, MIND at Home was successfully implemented in a diverse sample of 303 community-living individuals with memory disorders and was found to be acceptable to CGs, led to delays in time to transition from home, improved PWD quality of life, and CG time savings.

The current project is a 24-month, prospective, single- blind, parallel group, randomized controlled trial evaluating MIND-S in a cohort of 300 community-living PWD and their informal CGs in the Greater Baltimore area. Participants receiving MIND-S will get up to 18 months of care coordination by an interdisciplinary team comprised of trained memory care coordinators (non-clinical), a psychiatric nurse, and geriatric psychiatrist. The intervention involves 4 key components: identification of needs and individualized care planning (PWD and CG needs); dementia education and skill building; coordination, referral and linkage of services; and care monitoring.Participants in the comparison group will receive an initial in-home needs assessment and will be given the written results along with any recommendations for care that are indicated.

ELIGIBILITY:
Inclusion Criteria for PWD:

* Meets criteria for all-cause dementia using standard assessments and diagnostic criteria
* English speaking
* Has a reliable informal caregiver available and willing to participate
* Living at home the Greater Baltimore area

Exclusion Criteria:

* Planned move from home in less than 6 months
* On hospice or has end stage disease (bed-bound and non-communicative)
* Enrolled in another clinical trial for dementia or associated symptoms

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Time to long term care (LTC) placement or death | 18 months
  Time to long term care placement or death

SECONDARY OUTCOMES:
Cost-offset for total direct and indirect care costs | 18 months
  Estimates of cost-offset for the MIND-S program will be the cost-offset of MIND-S, defined as the net financial benefit of the program on total self-reported direct and indirect care costs. This will be calculated as the difference in the sum of all costs between MIND-S group and the sum of all costs in the augmented usual care from T1-T5 (baseline-18 months).
Cost-offset for total direct and indirect care costs | 24 months
  Estimates of cost-offset for the MIND-S program will be the cost-offset of MIND-S, defined as the net financial benefit of the program on total self-reported direct and indirect care costs. This will be calculated as the difference in the sum of all costs between MIND-S group and the sum of all costs in the augmented usual care from T1-T6 (baseline-24 months).
PWD unmet care needs | 18 months
  MIND at Home patient total unmet care needs as measured by the Johns Hopkins Dementia Care Needs Assessment 2.0 from baseline to 18 months compared to usual care group patient total unmet care needs from baseline to 18 months. (difference in slopes)
PWD unmet care needs | 24 months
  MIND at Home patient total unmet care needs as measured by the Johns Hopkins Dementia Care Needs Assessment 2.0 from baseline to 24 months compared to usual care group patient total unmet care needs from baseline to 24 months. (difference in slopes)
Neuropsychiatric symptoms (NPS) | 18 months
  MIND at Home patient Neuropsychiatric symptoms (NPS) as measured by the Neuropsychiatric Inventory-Questionnaire from baseline to 18 compared to usual care group patient NPS scores from baseline to 18 months. (difference in slopes)
Neuropsychiatric symptoms (NPS) | 24 months
  MIND at Home patient Neuropsychiatric symptoms (NPS) as measured by the Neuropsychiatric Inventory-Questionnaire from baseline to 24 compared to usual care group patient NPS scores from baseline to 24 months (difference in slopes)
Quality of life (QOL) | 18 months
  MIND at Home patient QOL as measured by the QOL-AD from baseline to 18 months compared to usual care group patient scores from baseline to 18 months (difference in slopes)
Quality of life (QOL) | 24 months
  MIND at Home patient QOL as measured by the QOL-AD from baseline to 24 months compared to usual care group patient scores from baseline to 24 months (difference in slopes)
Caregiver care unmet needs | 18 months
  MIND at Home caregiver total unmet care needs as measured by the Johns Hopkins Dementia Care Needs Assessment 2.0 from baseline to 18 months compared to usual care group patient total unmet care needs from baseline to 18 months. (difference in slopes)
Caregiver care unmet needs | 24 months
  MIND at Home caregiver total unmet care needs as measured by the Johns Hopkins Dementia Care Needs Assessment 2.0 from baseline to 24 months compared to usual care group patient total unmet care needs from baseline to 24 months. (difference in slopes)
Subjective caregiver burden | 18 months
  MIND at Home caregiver burden as measured by the Zarit Burden Interview from baseline to 18 months compared to usual care group patient burden from baseline to 18 months. (difference in slopes)
Subjective caregiver burden | 24 months
  MIND at Home caregiver burden as measured by the Zarit Burden Interview from baseline to 24 months compared to usual care group caregiver burden scores from baseline to 24 months. (difference in slopes)
Objective caregiver burden | 18 months
  MIND at Home caregiver burden as measured by time spent caregiving estimates from baseline to 18 months compared to usual care group time from baseline to 18 months. (difference in slopes)
Objective caregiver burden | 24 months
  MIND at Home caregiver burden as measured by time spent caregiving estimates from baseline to 24 months compared to usual care group time from baseline to 24 months. (difference in slopes)
Time to long term care (LTC) placement or death | 24 months
  Time to long term care placement or death

CONTACTS AND LOCATIONS:
Overall Officials: Quincy M Samus, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States